CLINICAL TRIAL: NCT02878772
Title: Vinpocetine Inhibits NF-κB-dependent Inflammation in Acute Ischemic Stroke
Brief Title: Vinpocetine Inhibits NF-κB-dependent Inflammation in Acute Ischemic Stroke Patients
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Tianjin Medical University General Hospital (Other)
Responsible Party: Principal Investigator, Junwei Hao, Professor, Tianjin Medical University General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TianjinMUGH1
Record Dates: First submitted 2016-08-04; First posted 2016-08-25 (Estimated); Last update posted 2016-08-25 (Estimated); Status verified 2016-08

CONDITIONS: Stroke; Immunoregulation; Inflammation; Vinpocetine
MeSH Terms: conditions — Stroke; Inflammation | interventions — vinpocetine; Aspirin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- vinpocetine group (Active Comparator): Aspirin, 10mg, po and 30 mg of the vinpocetine by intravenous infusion once daily, for fourteen consecutive days
  Interventions: Drug: vinpocetine; Drug: Aspirin
- Control group (Placebo Comparator): Patients will receive aspirin only.
  Interventions: Drug: Aspirin

INTERVENTIONS:
Drug: vinpocetine — 30 mg of the drug by intravenous infusion once daily, for fourteen consecutive days, beginning within one hour after the baseline MRI and no later than 48 hours after the onset of symptoms.
  Other Names: Cavinton
  Arms: vinpocetine group
Drug: Aspirin — 100mg, once daily, oral medication

SUMMARY:
Immunity and inflammation play critical roles in the pathogenesis of acute ischemic stroke. Therefore, immune intervention, as a new therapeutic strategy, is worthy of exploration. Here, investigators tested the inflammation modulator, vinpocetine, for its effect on the outcomes of stroke. For this multi-center study, investigators recruited 60 patients with anterior cerebral circulation occlusion and onset of stroke that had exceeded 4.5 hours but lasted less than 48 hours. These patients, after randomly division into two groups, received either standard management alone (controls) or standard management plus vinpocetine (30 mg per day intravenously for 14 consecutive days, Gedeon Richter Plc., Hungary).

ELIGIBILITY:
Inclusion Criteria:

* >18 years of age
* Anterior-circulation ischemic stroke: All patients had symptoms of focal neurological deficits and simultaneous radiological evidence (magnetic resonance imaging, MRI) of an ischemic brain lesion
* measurable neurological deficit (NIHSS > 5)
* interval between symptom onset and admission more than 4.5 hours and less than 48 hours. That is, all patients we recruited were beyond the 4.5 hours of symptom onset and, therefore, past the accepted time-window for thrombolytic therapy

Exclusion Criteria:

* hemorrhagic stroke and severe hemorrhage in other organs
* other diseases of the central nervous system (CNS)
* diabetes mellitus
* tumor or hematological systemic diseases
* any infection before acute ischemic stroke
* concomitant use of antineoplastic or immune modulating therapies
* contraindication to MRI

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-05; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
changes in lesion volume | lesion volume from baseline to day 7
  changes in lesion volume from baseline (DWI) to day 7 (Flair)
brain inflammatory level | day 7
  brain inflammatory level (MRS) at day 7
extent of clinical improvement | from baseline to day 7 and 14
  extent of clinical improvement at day 7 and 14, as measured by the changes on the NIHSS score from baseline to day 7 and 14

SECONDARY OUTCOMES:
probability of excellent recovery | at day 90
  probability of excellent recovery at day 90 (defined as a score of 0 or 1 on the mRS)
cytotoxic edema | day 3
  cytotoxic edema of day 3 (ADC value).

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Zhang F, Yan C, Wei C, Yao Y, Ma X, Gong Z, Liu S, Zang D, Chen J, Shi FD, Hao J. Vinpocetine Inhibits NF-kappaB-Dependent Inflammation in Acute Ischemic Stroke Patients. Transl Stroke Res. 2018 Apr;9(2):174-184. doi: 10.1007/s12975-017-0549-z. Epub 2017 Jul 9. PMID 28691141